CLINICAL TRIAL: NCT03845192
Title: Application and Validation of the New Oxygen Reserve Index in Infants < 2 Years Old
Brief Title: Oxygen Reserve Index for Kids
Acronym: ORIkids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Dr. Eva Wittenmeier:MD, principal investigator, Johannes Gutenberg University Mainz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ORIkids
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ORI measurement by Radical-97 (Other): In this arm ORI measurement is done from the beginning of the induction of anaesthesia until the end of the induction of anaesthesia or until the end of the stay in the operating theatre. The measurement to ORI is done by the "Radical-97" device by Masimo®
  Interventions: Device: ORI measurement by Radical 97

INTERVENTIONS:
Device: ORI measurement by Radical 97 — ORI measurement is done from the beginning of the induction of anaesthesia until the end of the induction of anaesthesia or until the end of the stay in the operating theatre. The measurement to ORI is done by the "Radical-97" device by Masimo®.

SUMMARY:
In infants less than two years old the new Oxygen Reserve Index (ORI) will be measured during general anaesthesia. It will evaluated if and how ORI-monitoring gives earlier warning of hypoxaemia than conventional oxygen saturation measurement.

DETAILED DESCRIPTION:
The Oxygen Reserve Index (ORI) is a new development in multiple wavelength pulse oximetry, reflecting the arterial partial oxygen pressure (PaO2) continuously and non-invasively by an index. In contrast to established standard oxygen saturation (SpO2) measurements, ORI detects a drop of PaO2 until the threshold of 100 mmHg. During anaesthesia induction-associated apnoeic periods ORI may detect a drop of PaO2 early enough for the anaesthesiologist to interrupt the intubation procedure and re-start oxygenation. In contrast, due to the flat upper part of the oxyhaemoglobin dissociation curve, SpO2 stays at values above 90% until PaO2 falls below 60mmHg. At this point, SpO2 drops rapidly and a pro- longed hypoxic dip is the consequence. To avoid this potentially harmful hypoxic dip, continuous monitoring of PaO2 using ORI would be advantageous during anaesthesia induction phase.

This clinical study aims to evaluate the time benefit between alarm of hypoxaemia by the ORI-monitoring and the start of the dropping of oxygen saturation. Pre-set and pre-described ORI-alarms will be checked for their utility and a new ORI-alarm will be defined that is potentially more useful. As secondary endpoints the study examines the correlation of ORI with PO2, the influence of patient or measurement characteristics on the correlation of ORI with PO2 and the influence of the measurement site on ORI-measurement.

ELIGIBILITY:
Inclusion Criteria:

* small infants < 2 years scheduled for elective surgery with general anaesthesia.

Exclusion Criteria:

* emergency procedures, lack of informed consent of legal guardian

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
time in seconds between ORI-dropping and dropping of SpO2 | during general anaesthesia of the infant
  Additionally a potential better definition of ORI-alarm than the preset or previously reported ORI-alarm will be defined

SECONDARY OUTCOMES:
correlation of ORI and PO2 | during general anaesthesia of the infant
influence of patient or measurement characteristics on the correlation of ORI and PO2 | during general anaesthesia of the infant
influence of measurement site on the correlation or ORI with PO2 and the influence of the measurement site on ORI measurement | during general anaesthesia of the infant

CONTACTS AND LOCATIONS:
Locations (1):
- Johannes Gutenbert University Centre, Mainz, Germany